CLINICAL TRIAL: NCT01288417
Title: Pharmacokinetic Study of the HCV Protease Inhibitor Boceprevir and the HIV Integrase Inhibitor Raltegravir
Acronym: OPAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 10.05
Record Dates: First submitted 2011-01-26; First posted 2011-02-02 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections; HCV Infections
Keywords: HIV infections; HCV infections; interaction; pharmacokinetics; raltegravir; boceprevir
MeSH Terms: conditions — HIV Infections | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- boceprevir + raltegravir (Experimental): 9 days of boceprevir 800mg TID; day 10 two doses of boceprevir 800mg and one dose of raltegravir 400mg
  Interventions: Drug: boceprevir; Drug: raltegravir
- raltegravir alone (Active Comparator): single dose of raltegravir 400mg
  Interventions: Drug: raltegravir

INTERVENTIONS:
Drug: boceprevir — 10 days of boceprevir 800mg TID
  Arms: boceprevir + raltegravir
Drug: raltegravir — raltegravir 400mg single dose
  Other Names: Isentress

SUMMARY:
The objective of this study is to evaluate the effect of boceprevir (steady state) on the pharmacokinetics of a single dose of raltegravir. The effect on the boceprevir pharmacokinetics of a single dose raltegravir will also be evaluated (compared to historical controls). Furthermore, the safety profile of the combination is studied.

DETAILED DESCRIPTION:
A considerable percentage of HIV infected patients is also infected with the hepatitis C virus (HCV). HIV/HCV co-infected patients are likely to simultaneously use treatment for their HIV infection as well as HCV treatment. Therefore, it is important to know if drug-drug interactions occur when combining those treatments.

Raltegravir is an HIV integrase inhibitor and approved by the FDA in 2007. Boceprevir is a potent HCV NS3 serine protease inhibitor and is currently in Phase III clinical development.

Combined use of boceprevir and raltegravir is not expected to give a major drug-drug interaction as raltegravir is not a CYP3A substrate and thus will not be affected by the strong inhibition of CYP3A by boceprevir. Raltegravir is metabolized by UGT but boceprevir is not known to influence UGT. However, recent data indicate that raltegravir is a P-gp substrate and boceprevir is a substrate and a moderate inhibitor of P-gp in vitro.

Even when no drug interaction is expected, it may be recommended to collect sufficient evidence that this is the case as in many cases un-expected drug-drug interactions have been observed in the past.

The current study is designed to evaluate the effect of steady state boceprevir on the pharmacokinetics of a single dose of raltegravir and the safety profile when used in combination. Furthermore the effect of a single dose raltegravir is studied on the pharmacokinetics of steady state boceprevir in comparison with historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years at scree-ning.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to the first dosing
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, haematology and urinalysis testing within 4 weeks prior to Day 1. Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges. If laboratory results are not within the reference ranges, the subject is included on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
* Subject has a normal blood pressure and pulse rate, according to the Investigator's judgement.

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Positive HIV test.
* Positive hepatitis B or C test.
* Pregnant female (as confirmed by an HCG test performed less than 4 weeks before Day 1) or breast-feeding female. Female subjects of childbearing potential without adequate contraception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the trial.
* Therapy with any drug (for two weeks preceding dosing), ex-cept for paracetamol.
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal and hepatic disorders, hormonal disorders (especially diabetes mellitus), coagulation disorders.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature and extent of the trial and the procedures required.
* Participation in a drug trial within 60 days prior to the first dose.
* Donation of blood within 60 days prior to the first dose.
* Febrile illness within 3 days before the first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
raltegravir concentrations | during 12hours on two occasions
  To determine the effect of chronic use of boceprevir on the single-dose pharmacokinetics of raltegravir 400mg in healthy volunteers

SECONDARY OUTCOMES:
adverse events | entire study
  to determine the safety of a single dose of raltegravir 400mg when combined with chronic use of boceprevir
boceprevir concentrations | during 8 hours on one occasion; predose 4 times over a period of 10 days
  To determine the effect of a single-dose pharmacokinetics of raltegravir 400mg on chronic use of boceprevir in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- CRCN, Nijmegen, Netherlands

REFERENCES:
- [Result] de Kanter CT, Blonk MI, Colbers AP, Schouwenberg BJ, Burger DM. Lack of a clinically significant drug-drug interaction in healthy volunteers between the hepatitis C virus protease inhibitor boceprevir and the HIV integrase inhibitor raltegravir. Clin Infect Dis. 2013 Jan;56(2):300-6. doi: 10.1093/cid/cis824. Epub 2012 Sep 21. PMID 23001704